CLINICAL TRIAL: NCT07369505
Title: A Phase 1b, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics of Sapu003 in Advanced mTOR-sensitive Solid Tumors (With or Without Exemestane)
Brief Title: Sapu003 in Advanced mTOR-sensitive Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SAPU NANO (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SP-03-B101
Record Dates: First submitted 2026-01-02; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Metastatic; Renal Cell Carcinoma (RCC); Neuroendocrine Tumors; Tuberous Sclerosis Complex (TSC); Hepatocellular Carcinoma (HCC)
Keywords: Sapu003; Everolimus for Injection; mTOR-Sensitive Solid Tumors; Renal Cell Carcinoma (RCC); Neuroendocrine Tumors (NETs); Tuberous Sclerosis Complex (TSC); Hepatocellular Carcinoma (HCC); everolimus; HR+/HER2-negative breast cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neuroendocrine Tumors; Tuberous Sclerosis; Carcinoma, Hepatocellular | interventions — Everolimus; Injections; exemestane

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b, open-label, sequential-assignment, dose-escalation study that uses a model-assisted Bayesian Optimal Interval (BOIN) design to guide intra-subject and inter-cohort dose decisions. Participants are enrolled in cohorts of three (with staggered "sentinel" dosing within each cohort) and receive once-weekly IV Sapu003 for four weeks per 28-day cycle. Two parallel disease-defined cohorts are studied:
  * Cohort A (HR+/HER2- breast cancer) - Sapu003 + daily oral exemestane
  * Cohort B (RCC, NETs, TSC-associated tumors, or HCC) - Sapu003 monotherapy
  Dose escalation proceeds from 5 mg/m² to 7.5 mg/m² to 10 mg/m² (with an optional -1 level of 3.5 mg/m²) according to BOIN escalation (λe ≈ 0.213) and de-escalation (λd ≈ 0.322) boundaries that target a DLT rate of 27 % during Cycle 1. Each dose level may expand to nine evaluable subjects; maximum sample size for the MTD determination is 27.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A - HR+/HER2- Breast Cancer (Experimental): Cohort A (Combination Therapy - HR+/HER2- Breast Cancer):
  Post-menopausal women with advanced or metastatic hormone-receptor-positive, HER2-negative breast cancer receive Sapu003 (everolimus for injection) as a 30-min IV infusion once weekly at 5, 7.5 or 10 mg/m², together with oral exemestane 25 mg once daily, repeated in 28-day cycles.
  Interventions: Drug: Sapu003; Drug: Exemestane 25 MG
- Cohort B - RCC / NET / TSC / HCC (Experimental): Cohort B (Monotherapy - RCC / NET / TSC / HCC):
  Adult patients with advanced renal cell carcinoma, neuro-endocrine tumours, tuberous-sclerosis-complex-associated tumours, or hepatocellular carcinoma receive Sapu003 (everolimus for injection) alone as a 30-min infusion once weekly at 5, 7.5 or 10 mg/m², repeated in 28-day cycles.
  Interventions: Drug: Sapu003

INTERVENTIONS:
Drug: Sapu003 — Sapu003 weekly IV at 5, 7.5 or 10 mg/m²
  Other Names: Sapu003/Everolimus for Injection
Drug: Exemestane 25 MG — Exemestane 25 mg QD (Breast Cancer Only)
  Other Names: Exemestane
  Arms: Cohort A - HR+/HER2- Breast Cancer

SUMMARY:
This is a phase 1b, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics of Sapu003 in combination with Exemestane in in patients with advanced mTOR-sensitive solid tumors (HR+/HER2-negative breast cancer, renal cell carcinoma [RCC], neuroendocrine tumors [NETs], tuberous sclerosis complex [TSC]-associated tumors, and hepatocellular carcinoma [HCC]).

DETAILED DESCRIPTION:
The study will include two cohorts:

* Cohort A: Patients with HR+/HER2-negative breast cancer who will receive Sapu003 in combination with exemestane.
* Cohort B: Patients with RCC, NETs, TSC-associated tumors, or HCC who will receive Sapu003 without exemestane.

The dose levels planned for this study are 5 mg/m², 7.5 mg/m², and 10 mg/m² administered as weekly 30-minute IV infusions, with each treatment cycle lasting 4 weeks (28 days).

The primary purpose of this study is to determine the maximum tolerated dose (MTD) of weekly intravenous Sapu003. Secondary objectives include characterizing the pharmacokinetic profile of Sapu003, evaluating its safety and tolerability, and assessing preliminary antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Sex and Age: Patients must be ≥ 18 years of age at the time of informed consent.

   * Cohort A (HR+/HER2- breast cancer): Eligible patients must be postmenopausal women, defined as women ≥ 18 years of age with amenorrhea for ≥ 12 consecutive months without another pathophysiological cause.
   * Cohort B (RCC, NETs, TSC-associated tumors, HCC): Eligible patients include both male and female adults with advanced disease.
2. Cohort A HR+/HER2- Breast Cancer:

   Eligible patients must meet all of the following:
   * Has histologically or cytologically documented advanced (metastatic or unresectable) hormone receptor-positive, HER2 negative breast cancer (advanced HR+ BC)
   * Has stage IV or locally advanced breast cancer per the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, Seventh Edition;
   * Has failed any combination endocrine therapy or relapse within 6 months of adjuvant chemotherapy for metastatic or locally advanced disease. Prior therapy should have included a non-steroidal aromatase inhibitor unless clinically contraindicated;
   * Has agreed to participate in the study and signed the informed consent form prior to participation in any study activities.
3. Cohort B Other Advanced mTOR-Sensitive Solid Tumors:

   Eligible patients must meet all of the following:
   * Has histologically or cytologically confirmed advanced (metastatic or unresectable) disease in one of the following tumor types:

     * Renal Cell Carcinoma (RCC)
     * Neuroendocrine Tumors (NETs)
     * Tuberous Sclerosis Complex (TSC)-associated tumors
     * Hepatocellular Carcinoma (HCC)
   * Has disease that is measurable and/or evaluable per RECIST v1.1 (or relevant criteria, if applicable).
   * Has progressed on or is intolerant to at least one prior line of standard therapy appropriate for the specific tumor type, unless no effective standard therapy exists.
   * Has agreed to participate in the study and signed the informed consent form prior to participation in any study activities.
4. Patients must be on stable doses of metformin or statin
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Life expectancy ≥ 3 months
7. Hematology/chemistry: Patient has adequate hematological, renal, and hepatic function as defined by the following Screening laboratory values obtained within 7 days prior to randomization and assessed based on local labs (patients should not have received a transfusion within 7 days before the Screening laboratory assessments):

   * Absolute neutrophil count (ANC) ≥ 2,000 cells/mm3 (2 x109/L)
   * Platelet count ≥ 100,000 cells/mm3 (100x109/L)
   * Hemoglobin≥ 9 g/dL
   * Serum creatinine≤ 1.5 x the upper limit of normal (ULN)
   * Total bilirubin ≤1.5 x ULN or direct bilirubin ≤1 x ULN for patients with total bilirubin levels > 1.5 ULN
   * AST (SGOT) / ALT (SGPT) ≤ 2.5 x ULN (≤5 x ULN for patients with metastases.)
   * GFR ≥ 50 mL/min/1.73m2 by the CKD-EPI or MDRD formulas.
8. All other clinical laboratory values deemed as normal or not clinically significant by the Principal Investigator/Sub-Investigator.
9. Breastfeeding: Patients must be non-lactating. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding must be discontinued prior to the first dose of study drug.
10. Female patients of reproductive potential to avoid becoming pregnant and to use effective contraception during the study and for 8 weeks after the last dose. Male patients with female partners of reproductive potential to use effective contraception during the study and for 4 weeks after the last dose.
11. Able and willing to adhere to all protocol requirements and study procedures throughout the course of the study.
12. Ability to comprehend and be informed of the nature of the study, as assessed by study clinic staff

Exclusion Criteria:

1. Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix, curatively treated in-situ carcinoma of the breast, or other solid tumors curatively treated with no evidence of disease for > 5 years.
2. Patients who have not completely recovered from any toxicities from previous chemotherapy, hormone therapy, immunotherapy, target therapy, or radiotherapies ≥ Grade 1 per NCI CTCAE version 5.0, with the exception of alopecia.
3. Patients who have received any of the following treatments within the specified timeframes prior to screening:

   * Prior chemotherapy within 30 days prior to screening (42 days for mitomycin C or nitrosoureas).
   * Prior immunotherapy, prior anti-tumor hormonal therapy (for breast cancer patients), and prior radiotherapy within 30 days prior to screening.
   * Radiotherapy is not allowed during study. Administration of other chemotherapy, immunotherapy, or anti-tumor hormonal therapy during the study is not allowed.
4. Patients had major surgery within 30 days prior to randomization, or patients have not recovered from prior major surgery.
5. Sensory / Peripheral neuropathy of > Grade 1 per NCI CTCAE version 5.0 at Screening.
6. Patients with active brain metastases. Patients with treated brain metastases are eligible provided they have no evidence of active brain disease and are off of definitive therapy (including steroids) at least 3 months prior to randomization.
7. Known history or presence of any clinically significant disease or condition other than cancer unless determined as not clinically significant by the Principal Investigator/Sub-Investigator. This includes, but is not limited to, the following: hepatic, renal/genitourinary, gastrointestinal (e.g., intra-abdominal inflammation), cardiovascular (e.g., congestive heart failure, ventricular arrhythmia, myocardial infarction, unstable angina pectoris), cerebrovascular, pulmonary (e.g., interstitial lung disease), endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological, or hematological (e.g., bleeding diathesis or coagulopathy).
8. History of difficulty with donating blood or difficulty in accessibility of central line.
9. Known history or presence of:

   * Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C (serology to confirm absence is required within 7 days prior to randomization and assessed based on local labs);
   * Alcohol abuse or dependence within one year prior to randomization;
   * Drug abuse or dependence (marijuana, amphetamines, barbiturates, cocaine, opiates and benzodiazepines);
   * Hypersensitivity or idiosyncratic reaction to everolimus, other rapamycin derivatives or its excipients
   * Severe allergic reactions (e.g., anaphylactic reactions, angioedema).
10. Patients may not participate in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or the use of investigational devices with therapeutic intent within 30 days prior to randomization and while enrolled in this study. Caution is recommended when administering Sapu003 and concomitantly with known substrates, PgP inhibitors, inhibitors, and inducers of the cytochrome P450 isoenzymes CYP2C8 and CYP3A4.
11. Use of any strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates (phenobarbital), carbamazepine, phenytoin and rifampin), in the previous 14 days before randomization until the last blood draw in the study.
12. Acute active infection requiring antibiotics, antiviral agents, or antifungal agents within 14 days prior to randomization
13. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose Limiting Toxicities (DLTs) of Sapu003 in Patients with Advanced mTOR-Sensitive Solid Tumors | The primary outcome timeframe is assessed during the first 28-day cycle of treatment, specifically looking at dose-limiting toxicities (DLTs) to determine the maximum tolerated dose (MTD) of Sapu003
  The primary outcome of the study is to determine the Maximum Tolerated Dose (MTD) of Sapu003, defined as the dose level where the estimated true probability of Dose-Limiting Toxicity (DLT) is closest to the target toxicity probability (TTP) of 0.27. This will be evaluated through a dose-escalation design, where patients receive Sapu003 intravenously every week, with doses ranging from 5 to 10 mg/m². The analysis will include the cumulative number of DLTs observed at each dose level, guiding decisions for dose escalation or de-escalation, ultimately reporting the recommended MTD based on isotonic regression estimates

SECONDARY OUTCOMES:
Pharmacokinetic Endpoint - Cmax | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Peak Plasma Concentration (Cmax)
Pharmacokinetic Endpoint - AUClast | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Area Under the Curve from time zero to the last quantifiable concentration (AUClast)
Pharmacokinetic Endpoint - AUCinf | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Area Under the Curve to Infinity (AUCinf)
Pharmacokinetic Endpoint - tmax | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Time to reach maximum concentration (tmax)
Characterization of the Pharmacokinetic Endpoint - t1/2 | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Elimination half-life (t1/2)
Pharmacokinetic Endpoint - CL | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Clearance (CL)
Pharmacokinetic Endpoint - Vd | Week 1 of Cycle 1 and Cycle 2 (28 days per Treatment Cycle)
  Characterization of the Pharmacokinetic Endpoint - Volume of Distribution (Vd)
Anti-Tumor Activity Assessment - ORR | Through study completion
  Preliminary anti-tumor activity - ORR (Objective Response Rate)
Anti-Tumor Activity Assessment - DCR | Through study completion
  Preliminary anti-tumor activity - DCR (Disease Control Rate)
Anti-Tumor Activity Assessment - PFS | Until the end of the study
  Preliminary anti-tumor activity - PFS (Progression-Free Survival)
Anti-Tumor Activity Assessment - DoR | Until the end of the study
  Preliminary anti-tumor activity - DoR (Duration of Response)
Anti-Tumor Activity Assessment - OS | Until the end of the study
  Preliminary anti-tumor activity - OS (Overall Survival)

CONTACTS AND LOCATIONS:
Locations (1):
- SOCRU, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No